CLINICAL TRIAL: NCT01027312
Title: Reproducibility and Clinical Usefulness of AARV (Assessment of Ability Related to Vision)
Brief Title: Assessment of Ability Related to Vision
Acronym: AARV
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal Investigator, Wills Eye
Other Study IDs: IRB#07-842
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; quality of life; daily living activities; visual fields; contrast sensitivity
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma Patients: Glaucoma patients covering the entire range of visual field loss from none to advanced.
- Control Group: Aged matched people with no eye diseases.

SUMMARY:
To determine the clinical usefulness of a refined third-generation instrument - The Assessment of Ability Related to Vision (AARV) in establishing the amount of disability, charting the detrimental effects of progressive disease and establishing the beneficial effects of treatment

DETAILED DESCRIPTION:
This research study is designed to test the usefulness and repeatability of testing how much disability is caused by vision loss due to glaucoma. We are recruiting 100 patients with glaucoma and 20 healthy (have no eye disease) individuals to be enrolled in this study. The healthy study participants will be enrolled in order to describe how a healthy individual will perform on the test designed to assess one's performance when completing ten activities of daily living.

Clinical testing will be conducted by binocular and monocular visual fields, contrast sensitivity and visual acuity. The NEI-VFQ 15 Quality of Life Questionnaire will be used to measure patients perception of how well they are doing.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 yrs of age and older
* must understand and respond to spoken English and be fully literate.

Exclusion Criteria:

* Patients with significant neurological problems (like Parkinson's disease), motor problems (like arthritis) or other significant illnesses that may prevent them from completing the testing involved in the study (like advanced heart failure).
* Patients who have received training related to low vision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred patients with bilateral unstable glaucoma and twenty patients who appear to be normal will be enrolled.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
the reproducibility of AARV, and its relationship to standard clinical tests | Day 1, 1 week, 6 months, 1 year

SECONDARY OUTCOMES:
A better estimate of the reproducibility of standard clinical tests. | Day 1, 1 week, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Wills Eye Institute

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been written and published

REFERENCES:
- [Result] Wei H, Sawchyn AK, Myers JS, Katz LJ, Moster MR, Wizov SS, Steele M, Lo D, Spaeth GL. A clinical method to assess the effect of visual loss on the ability to perform activities of daily living. Br J Ophthalmol. 2012 May;96(5):735-41. doi: 10.1136/bjophthalmol-2011-300093. Epub 2012 Jan 12. PMID 22241927